CLINICAL TRIAL: NCT05291689
Title: A Phase 2a, Open-label, Single-arm Study to Evaluate the Efficacy, Safety, and Tolerability of MORF-057 in Adults With Moderately to Severely Active Ulcerative Colitis (EMERALD-1)
Brief Title: A Phase 2a Open-Label Study to Evaluate the Efficacy and Safety of MORF-057 in Adults With UC
Acronym: EMERALD-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Morphic Therapeutic, Inc. (A Wholly Owned Subsidiary of Eli Lilly and Company) (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27506; J6E-MC-KWAL (Other: Eli Lilly and Company); MORF-057-201 (Other: Morphic Therapeutic, Inc)
Record Dates: First submitted 2022-03-10; First posted 2022-03-23 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Bowel Diseases; Colitis, Ulcerative
Keywords: Ulcerative Colitis (UC); Inflammatory Bowel Disease (IBD); a4b7; Moderately to severely active ulcerative colitis; Integrin
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MORF-057 (Experimental)
  Interventions: Drug: MORF-057

INTERVENTIONS:
Drug: MORF-057 — MORF-057 is a small molecule that is designed to selectively inhibit integrin α4β7 and is administered orally.

SUMMARY:
This is an open-label, single arm, multicenter, Phase 2a study evaluating the efficacy, safety, and tolerability of MORF-057 in adult patients with Moderately to Severely Active Ulcerative Colitis (UC)

DETAILED DESCRIPTION:
The main part of this Phase 2a study will consist of 3 study periods: a Screening Period, a Treatment Period and a Safety Follow-up Period. All participants who complete the open-label Treatment Period will have the opportunity to continue their treatment in an optional 26-week Long-term Extension study after completing the Week 52 assessments.

ELIGIBILITY:
Inclusion Criteria:

* Has signs/symptoms of moderately to severely active UC for at least 3 months prior to Screening
* Has evidence of UC extending at least 15 cm from the anal verge
* Is bio-naïve or had an inadequate response, loss of response, or intolerance to other UC drugs
* Agrees to abide by the study guidelines and requirements
* Capable of giving signed informed consent

Exclusion Criteria:

* Diagnosed with indeterminate colitis, microscopic colitis, ischemic colitis, radiation colitis, or Crohn's disease or has clinical findings suggestive of Crohn's disease
* Has positive findings on a subjective neurological screening questionnaire
* Has a concurrent, clinically significant, serious, unstable comorbidity
* Primary non-responder to vedolizumab or other integrin inhibitors
* Participation in any other interventional study or received any investigational therapy within 30 days
* Previous exposure to MORF-057 and/or a known hypersensitivity to drugs with a similar mechanism to MORF-057
* Unable to attend study visits or comply with study procedures

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2025-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (5):
  - Clinical Study Site, Tampa, Florida
  - Clinical Study Site, Lafayette, Louisiana
  - Clinical Study Site, Freehold, New Jersey
  - Clinical Study Site, Brooklyn, New York
  - Clinical Study Site, New York, New York
- Poland (10):
  - Clinical Study Site, Bydgoszcz
  - Clinical Study Site, Elblag
  - Clinical Study Site, Katowice
  - Clinical Study Site, Lodz
  - Clinical Study Site, Oświęcim
  - Clinical Study Site, Sopot
  - Clinical Study Site, Sosnowiec
  - Clinical Study Site, Staszów
  - Clinical Study Site, Tychy
  - Clinical Study Site, Warsaw

REFERENCES:
- [Derived] Sands BE, Schreiber S, Danese S, Kierkus J, Abhyankar B, Choi MY, Soo C, Wu Y, Sun F, Lee D, Cui D, Mangada M, Singhal P, Hussain A, Rogers BN, Peyrin-Biroulet L, Feagan BG. A Phase 2 Study of MORF-057, an Oral alpha4beta7 Integrin Inhibitor in Moderately to Severely Active Ulcerative Colitis. Clin Gastroenterol Hepatol. 2025 Aug 6:S1542-3565(25)00648-2. doi: 10.1016/j.cgh.2025.07.030. Online ahead of print. PMID 40769468

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MORF-057
Started | 35
Completed | 18
Not Completed | 17
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 10
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | MORF-057
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 33
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
  Poland | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Robarts Histopathology Index (RHI) Score
Description: Robarts Histopathology Index (RHI) Score: the total RHI Score ranges from 0 (no disease activity) to 33 (severe disease activity)
Time Frame: From baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MORF-057
Number analyzed (Participants) | 35
score on a scale | -6.4 (11.18)

2. Secondary Outcome: Change From Baseline to Week 12 in the Modified Mayo Clinic Score
Description: The Modified Mayo Clinic Score (mMCS) is a composite of the following Mayo Clinic Score subscores: Endoscopy subscore (range: 0=Normal or inactive disease to 3=Severe disease (spontaneous bleeding, ulceration), Stool Frequency subscore (range: 0=Normal number of stools for this participant to 3=5 or more stools more than normal), and Rectal Bleeding subscore (range: 0=No blood seen to 3=Blood alone passed).
  The total mMCS ranges from 0 to 9, with higher scores indicating more severe disease.
Time Frame: From baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MORF-057
Number analyzed (Participants) | 35
score on a scale | -2.3 (2.14)

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) During Multiple Doses of MORF-057
Description: To determine the Maximum Plasma Concentration of MORF-057, blood samples were collected per the study protocol at the following time points: Study Day 1 (first dose), predose and 1, 2, 3, 4, and 6 hours post the AM dose; Week 2, predose and 1, 2, 3, 4, and 6 hours post the AM dose; Week 6, predose and 1 and 3 hours post the AM dose; Week 12, predose and 1, 2, 3, 4, and 6 hours post the AM dose. On Study Day 1, Week 2, and Week 12, blood sampling for pharmacokinetics was optional at 8, 10, and 12 hours post the AM dose.
Time Frame: 12 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MORF-057
Number analyzed (Participants) | 28
ng/mL | 766 (46.4)

4. Secondary Outcome: Time to Reach Cmax (Tmax) During Multiple Doses of MORF-057
Description: To determine the Tmax of MORF-057, blood samples were collected per the study protocol at the following time points: Study Day 1 (first dose), predose and 1, 2, 3, 4, and 6 hours post the AM dose; Week 2, predose and 1, 2, 3, 4, and 6 hours post the AM dose; Week 6, predose and 1 and 3 hours post the AM dose; Week 12, predose and 1, 2, 3, 4, and 6 hours post the AM dose. On Study Day 1, Week 2, and Week 12, blood sampling for pharmacokinetics was optional at 8, 10, and 12 hours post the AM dose.
Time Frame: 12 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | MORF-057
Number analyzed (Participants) | 28
hours | 2.014 (58.4534)

5. Secondary Outcome: Area Under the Curve (AUC) Following Multiple Doses of MORF-057
Description: To determine the area under the concentration-time curve of MORF-057, blood samples were collected per the study protocol at the following time points: Study Day 1 (first dose), predose and 1, 2, 3, 4, and 6 hours post the AM dose; Week 2, predose and 1, 2, 3, 4, and 6 hours post the AM dose; Week 6, predose and 1 and 3 hours post the AM dose; Week 12, predose and 1, 2, 3, 4, and 6 hours post the AM dose. On Study Day 1, Week 2, and Week 12, blood sampling for pharmacokinetics was optional at 8, 10, and 12 hours post the AM dose.
Time Frame: 12 weeks
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | MORF-057
Number analyzed (Participants) | 27
hours*ng/mL | 3070 (45.7)

ADVERSE EVENTS:
Time Frame: 52-week treatment period
Description: Adverse events will be reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative).
  The Investigator and any qualified designees are responsible for detecting, documenting, and recording events that meet the definition of an AE or SAE. For each AE, the Investigator will evaluate and report the onset, resolution, severity, causality, action taken, outcomes, and whether or not it caused the participant to discontinue.
Arm/Group | MORF-057
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 18/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MORF-057 (N=35)
Colitis ulcerative (Gastrointestinal disorders) | 7
Anal fistula (Gastrointestinal disorders) | 2
Nasopharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Viral upper respiratory tract infection (Infections and infestations) | 2
Anaemia (Blood and lymphatic system disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per the study protocol: "The results of this study may be published or presented at scientific meetings. If this is foreseen, the Investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission."

DOCUMENTS (2):
  • Study Protocol (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT05291689/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT05291689/SAP_001.pdf